CLINICAL TRIAL: NCT04360837
Title: PEEP Incremental and Decremental Alveolar Recruitment of Critically Ill COVID-19 Patients Under Electric Impedance Tomography (EIT)
Brief Title: PEEP Incremental and Decremental Alveolar Recruitment of Critically Ill Corona Virus Disease-19 (COVID-19) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Collaborators: Hochschule Furtwangen University (Other); Budapest University of Technology and Economics (Other)
Responsible Party: Principal Investigator, András Lovas, consultatnt in critical care and anaesthesiology, Szeged University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVID-19EIT
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Virus; Pneumonia; Atelectasis
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEP incremental-decremental alveolar recruitment (Experimental): 1. installing EIT belt over the chest at the level of the 5th intercostal space and adjustment of the default recruitment settings in pressure control ventilation mode: pressure control 15 cmH20, PEEP 10 cmH2O, fraction of inspired oxygen (FiO2) and respiratory rate according to the discretion of the attending physician, recording basal parameters
  2. implementation of recruitment:
     * increment phase: increasing PEEP by 3 cmH2O in every two minutes from 10 cmH2O until top of PEEP 25 cmH2O
     * decrement phase: decreasing PEEP by 3 cmH20 in every two minutes from 25 cmH20 until the basal PEEP 10 cmH20
     * end inspiratory hold manoeuvre at every PEEP level
  3. recording closing parameters
  Repeating the above detailed intervention once daily as long as the patient is controlled ventilation.
  Interventions: Procedure: alveolar recruitment

INTERVENTIONS:
Procedure: alveolar recruitment — incremental and decremental positive end-expiratory pressure alveolar recruitment

SUMMARY:
COVID-19 originated from Severe Acut Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) infection leads to critical condition due to hypoxemic respiratory failure with the background of viral pneumonia. Both alevolar recruitment and the subsequent optimal positive end-expiratory pressure (PEEP) adjustment has a pivotal role in the elimination of atelectasis developed by inflammation in the lung parenchyma The gold standard of the follow up of recruitment manoeuvre is the chest computed tomography (CT) examination. However, reduction of intrahospital transport and the exposure with healthcare workers are recommended because of the extremely virulent pathogen spreading easily by droplet infection. In this case bedside investigations have an utmost importance in the management of hygiene regulations.

Electric impedance tomography (EIT) is a non-invasive, radiation free functional imaging technique easily applicable at the bedside.

DETAILED DESCRIPTION:
COVID-19 originated from Severe Acut Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) infection leads to critical condition in 5% of the cases due to hypoxemic respiratory failure with the background of viral pneumonia. 90% of these patients require invasive mechanical ventilation on critical care units. Both alevolar recruitment and the subsequent optimal positive end-expiratory pressure (PEEP) adjustment has a pivotal role in the eliminitaion of atelectasis developed by inflammation in the lung parenchyma.

The gold standard of the follow up of recruitment manoeuvre is the chest computed tomography (CT) examination. However, reduction of intrahospital transport and the exposure with healthcare workers are recommended because of the extremely virulent pathogen spreading easily by droplet infection. In this case bedside investigations have an utmost importance in the management of hygiene regulations.

Electric impedance tomography (EIT) is a non-invasive, radiation free functional imaging technique easily applicable at the bedside. With the help of EIT, intrathoracic impedance changes, resulting from air and blood volume variations, can be determined by circumferentially attached surface electrodes around the thorax, applying small alternating currents and measuring differences in surface potentials. The calculated difference in potential is utilised to reconstruct impedance images what is employed to assess ventilation and perfusion distribution. Several local and global variances can be estimated just like the ratio fo atelectatic/overdistended alveoli, the ratio of aeration in the anterior/posterior regions, the inhomogeneity of aeration or regional compliance.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 positivity confirmed by polymerase chain reaction
* orotracheally intubated patients
* pressure control ventilation mode
* sedation level of minimum -4 on the Richmond Agitation Sedation Scale (RASS)

Exclusion Criteria:

* age under 18
* pregnancy
* pulmonectomy, lung resection in the past medical history
* clinically end stage chronic obstructive pulmonary disease
* sever hemodynamic instability (vasopressor refractory shock)
* sever bullous emphysema and/or spontaneous pneumothorax in the past medical history chest drainage in situ due to pneumothorax and/or bronchopleural fistula

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in lung compliance | 20 minutes
  Estimation of change in compliance (ml/cmH2O) from the beginning to end of of the incremental/decremental PEEP alveolar recruitment.
Change in global impedance | 20 minutes
  Estimation of change in global impedance (%) from the beginning to end of of the incremental/decremental PEEP alveolar recruitment.
Change in recruitability | 7 days
  Estimation of change in global impedance (%) on a daily manner.

SECONDARY OUTCOMES:
Gas exchange | 20 minutes and 7 days
  Change in arterial partial pressure of oxygen (PaO2) (mmHg) following recruitment
Plateau pressure | 20 minutes and 7 days
  Change in plateau pressure (cmH2O) following recruitment
End expiratory lung impedance (EELI) | 20 minutes and 7 days
  Change in end expiratory lung impedance (%)
Antero-to-posterior ventilation ratio | 20 minutes and 7 days
  Change in antero-to-posterior ventilation ratio (%) following intervention
Center of ventilation | 20 minutes and 7 days
  Change in center of ventilation (%) following intervention
Global inhomogeneity index | 20 minutes and 7 days
  Change in global inhomogeneity index (%) following intervention

CONTACTS AND LOCATIONS:
Overall Officials: András Lovas, MD PhD, Principal Investigator — SZTE AITI
Locations (1):
- University of Szeged, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gattinoni L, Caironi P, Cressoni M, Chiumello D, Ranieri VM, Quintel M, Russo S, Patroniti N, Cornejo R, Bugedo G. Lung recruitment in patients with the acute respiratory distress syndrome. N Engl J Med. 2006 Apr 27;354(17):1775-86. doi: 10.1056/NEJMoa052052. PMID 16641394
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Background] Lovas A, Hankovszky P, Korsos A, Kupcsulik S, Molnar T, Szabo Z, Babik B. [Importance of the imaging techniques in the management of COVID-19-infected patients]. Orv Hetil. 2020 Apr 1;161(17):672-677. doi: 10.1556/650.2020.31814. Hungarian. PMID 32324360
- [Result] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Derived] Lovas A, Chen R, Molnar T, Benyo B, Szlavecz A, Hawchar F, Kruger-Ziolek S, Moller K. Differentiating Phenotypes of Coronavirus Disease-2019 Pneumonia by Electric Impedance Tomography. Front Med (Lausanne). 2022 May 19;9:747570. doi: 10.3389/fmed.2022.747570. eCollection 2022. PMID 35665323